CLINICAL TRIAL: NCT06517030
Title: Clinical and Radiographic Evaluation of a Socket Reconstruction Technique and Immediate Implant Placement With Two Different Bone Substitute Materials: a Multicentric Randomized Clinical Trial.
Brief Title: Socket Reconstruction Technique and Immediate Implant Placement With Two Different Bone Substitute Materials.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo de Sanctis, Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Botiss-1
Record Dates: First submitted 2024-03-06; First posted 2024-07-24 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Intervention Model Description: The present research is a national multicentric prospective parallel double-blinded (both the patient and the investigator who will perform the measurements are blind) randomized controlled clinical trial. It is a superiority comparative study on a medical device CE marking, used according to the intended use subject to the CE marking.
Who Masked: Participant, Outcomes Assessor
Masking Description: A randomization list will be generated in blocks: patients will be divided in 3 blocks according to the study center and the treatment will be assigned at random in each block to ensure a balanced distribution of the tested interventions, with a ratio test:control=1:1. The investigator who will generate the allocation sequence will not be the person who will determine eligibility and entry of patients. The assignments (A or B group) will enclose in serially numbered, opaque, sealed envelopes, each bearing on the outside only the letter corresponding to the name of the center (M, B, S) and a number (from 1 to 10).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (DBBM+HA) (Experimental): In Test group, the gap between the implant surface and the bone plates will be filled with deproteinized bovine bone mineral with hyaluronic acid (Botiss Cerabone Plus; Botiss biomaterials, Hauptstr. 28 15806 Zossen, Germany). The material will be pre-wetted in saline, inserted in the gap and once soaked in blood, it will be gently pressed to the bone walls to completely fill the space and around buccal aspects of the exposed implant surface, up to the top of the abutment.
  Interventions: Procedure: Tooth Extraction; Procedure: Immediate Implant Placement; Procedure: Socket reconstruction with DBBB+HA; Procedure: CTG placement
- Control group (DBBM) (Active Comparator): In Control group, deproteinized bovine bone mineral (DBBM) (Bio-Oss Collagen; Geistlich Pharma, Wolhusen, Switzerland) will be positioned in the gap. The material will be pre-wetted in saline, inserted in the gap and once soaked in blood, it will be gently pressed to the bone walls to completely fill the space and around buccal aspects of the exposed implant surface, up to the top of the abutment.
  Interventions: Procedure: Tooth Extraction; Procedure: Immediate Implant Placement; Procedure: Socket reconstruction with DBBB; Procedure: CTG placement

INTERVENTIONS:
Procedure: Tooth Extraction — After local anaesthesia, a buccal split-full-split-thickness envelope flap will be elevated, and the tooth will be extracted a-traumatically.
Procedure: Immediate Implant Placement — After providing that the extraction socket will meet the inclusion criteria, an implant will be immediately inserted with 1 mm of its transmucosal portion positioned under the interproximal bone crest.
Procedure: Socket reconstruction with DBBB+HA — The gap between the implant surface and the bone plates will be filled with deproteinized bovine bone mineral with hyaluronic acid (DBBM+HA).
  Arms: Test group (DBBM+HA)
Procedure: Socket reconstruction with DBBB — The gap between the implant surface and the bone plates will be filled with deproteinized bovine bone mineral (DBBM).
  Arms: Control group (DBBM)
Procedure: CTG placement — Once the appropriate healing abutments will be installed, a CTG will be utilized as a barrier membrane. Then, the buccal flap will be coronally advanced and will be adapted to the healing abutment.

SUMMARY:
The present research is a national multicentric prospective parallel double-blinded (both the patient and the examiner are blind) randomized controlled clinical trial. It is a superiority comparative study on a medical device CE (conformité européenne) marking, used according to the intended use subject to the CE marking.

The hypothesis tested is: the socket reconstruction procedure performed in conjunction with Immediate implant placement (IIP) with the use of Deproteinized bovine bone mineral + hyaluronic acid (DBBM+HA, Cerabone plus) leads to a greater increase in the vertical buccal bone height than same procedure with deproteinized bovine bone mineral alone (DBBM, Bio-oss Collagen).

DETAILED DESCRIPTION:
The present research is a national multicentric prospective parallel double-blinded (both the patient and the investigator who will perform the measurements are blind) randomized controlled clinical trial. It is a superiority comparative study on a medical device CE marking, used according to the intended use subject to the CE marking.

The hypothesis tested is: the socket reconstruction procedure performed in conjunction with IIP with the use of DBBM+HA leads to a greater increase in the vertical buccal bone height than same procedure with DBBM alone.

The present study will be reported according to the CONSORT statement for improving the quality of reports of parallel-group randomized trials (http://www.consort-statement.org/).

Patients will be randomly treated by means of IIP+connective tissue graft (CTG)+DBBM+HA (Test group or A group) or IIP+CTG+DBBM (Control group or B group). A randomization list will be generated in blocks: patients will be divided in 3 blocks according to the study center (M=San Raffaele Hospital, Milan; B=University of Bologna; S=University of Siena) and the treatment will be assigned at random in each block to ensure a balanced distribution of the tested interventions, with a ratio test:control=1:1. The investigator who will generate the allocation sequence will not be the person who will determine eligibility and entry of patients. The assignments (A or B group) will enclose in serially numbered, opaque, sealed envelopes, each bearing on the outside only the letter corresponding to the name of the center (M, B, S) and a number (from 1 to 10). A designated investigator for each center will be responsible to ensure that the envelopes will be opened sequentially, and only after the patient will undergo extraction of the hopeless tooth, implant placement, and clinical measurement assessment. For each patient, a sequential number will be assigned based on the date of enrollment, and the envelope with the corresponding number will be opened for each of them.

Both the investigator who will perform the measurements and the patients will be blinded to the randomization. The principal investigator (PI) will make sure patients are blind by simply not telling them there is a difference between the two medical devices; while he will ensure that investigator (who will perform the measurements) is blind by assigning a code or an identifying number to the two treatment groups so that they cannot know which device has been used.

Patients will be followed for 6 months after surgery.

The undermentioned 5 follow-up visits, which are standard of practice for all implant-bearing patients, will be scheduled for each patient for both treatment groups at:

1. 7±2 days post-surgery - clinical and photographic examination, collection of VAS (Visual Analogue Scale).
2. 14±4 days post-surgery - suture removal, clinical and photographic examination.
3. 1 month±7 days post-surgery - clinical and photographic examination.
4. 3 months±5 days post-surgery - clinical and photographic examination, measurements of the following parameters: Gingival recession depth (REC in mm), Keratinized tissue width (KTW in mm), Soft tissue thickness (GT in mm), Pocket probing depth (PPD in mm), Bleeding on probing (BoP), Plaque index (PI).
5. 6 months ±1 month post-surgery - clinical and photographic examination, CBCT scan, periapical radiography, 3D digital dental impression, measurements of the following parameters: Gingival recession depth (REC in mm), Keratinized tissue width (KTW in mm), Pocket probing depth (PPD in mm), Bleeding on probing (BoP), Plaque index (PI).

After the visit at 6 months, each patient will then be considered "off study" (e.g. subject has completed treatment and all follow-up visits).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the trial.
2. In good general health as evidenced by medical history.
3. Presenting a single hopeless tooth candidate for extraction in the maxillary or mandibular area (from second premolar to second premolar, intercalated or the last tooth of dental arch) in need of a single implant-supported fixed prosthetic rehabilitation.
4. Presence of >3mm of buccal wall dehiscence evaluated using Cone Beam Computed Tomography (CBCT).
5. In healthy periodontal conditions (i.e., no presence of sites ≥ 4 mm and/or presence of intra-bony defects in the selected sites, full mouth plaque score < 20% and full-mouth bleeding score < 20%).

Exclusion Criteria:

1. Current or previous use of immunosuppressant, bisphosphonate, or high-dose corticosteroid therapy.
2. Presence of inflammatory and autoimmune disease of the oral cavity.
3. Severe or poorly controlled diabetes or previous radiotherapy of head area.
4. Contraindications to dental and/or surgical interventions (e.g. severe endocrine bone diseases, severe metabolic bone disorders, malignant tumour diseases).
5. Individuals who are smokers of >10 cigarettes/day.
6. Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
7. Presence of <3mm of dehiscence of buccal walls of the socket after tooth extraction.
8. Presence of a distance between the interdental bone crest and buccal bone crest <3 mm after tooth extraction.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Vertical buccal bone height changes (∆VBBH). | at baseline and at 6 months after procedure
  the vertical linear distance from point A (the most coronal point of the buccal crest of the baseline socket) to point B (the most coronal point of the buccal crest at 6 months after implant insertion)

SECONDARY OUTCOMES:
Width of keratinized tissue (KTW). | at baseline and at 6 months after treatment.
  Measured at the buccal aspect, as the distance between gingival margin and mucogingival junction.
Soft tissue contour changes. | at baseline and at 6 months after treatment.
  Linear and volumetric measurements will be performed using Stl files superimposition.
Soft tissue thickness (STT). | at baseline and at 6 months after treatment.
  Superimposition of DICOM file, representing hard tissue volume, to STL file representing soft tissue contour, will be used to measure the buccal soft tissue thickness in the two different treatment groups.
Horizontal Buccal Bone Changes. | at baseline and at 6 months after treatment.
  The horizontal linear distance between the outer surface of buccal bone at baseline and that at 6 months will be evaluated.
Osseous Ridge Width Changes. | at baseline and at 6 months after treatment.
  the horizontal linear distance from the outer surface of buccal bone to the outer surface of palatal/lingual bone, measured at baseline and at 6 months. The osseous ridge width changes in millimetres (mm) and in percentage (%ORR) will be also calculated.
Wound healing index (WHI). | at 7 and 14 days after treatment.
  The following criteria will be used:
  * score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort or flap dehiscence + intact papillae height
  * score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration + reduced papillae height
  * score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration + loss of papillae height
Post-surgical pain (PP) | at 7 and 14 days after treatment.
  Subjects will be also asked to evaluate pain perception at day 7 and day 14 using a visual analogue scale (VAS) score (0 = no pain 10 = maximal pain).
Amount of drug intake | from the day of surgery until day 14
  The daily consumption of analgesics/anti-inflammatory medications from the day of surgery until day 14 will be calculated.
Handling of materials. | at the day of the surgery
  The clinical handling of the two grafts will be assessed retrospectively by the surgeons using a visual analogue scale (VAS, 0 = easy to be applied, 10 = very difficult to be applied)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No